CLINICAL TRIAL: NCT00603057
Title: Using Functional Image and Circulating Molecular Markers to Predict Tumor Response and Lung Toxicity in Treatment of Lung Cancer
Brief Title: Using Imaging and Molecular Markers to Predict Tumor Response and Lung Toxicity in Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2006.040; HUM00002913 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2008-01-04; First posted 2008-01-28 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung Cancer Imaging Patients: Adult patients (>18 years of age)with histologically confirmed or clinically diagnosed lung cancer who require radiation therapy, with or without surgery and with or without chemotherapy.

SUMMARY:
Successful treatment of non-small cell lung cancer with radiation therapy requires that the physicians determine exactly where the tumor is in your body and protect your normal tissue. This study is designed to apply functional imaging, Fluorodeoxyglucose-Positron Emission Tomography (FDG-PET) and Ventilation/Perfusion Single Photon Emission Computerized Tomography (V/Q SPECT), before treatment and then again during treatment to see if it helps predict how well the treatment works for your cancer and how well your lung functions during treatment. A Computerized Tomography (CT) will also be performed along with both of these procedures to help the researchers see clearly where your cancer or your healthy lung is located.

The researchers are also doing blood tests in this study to look for markers in your blood and to see if it helps them in determining your risk of developing side effects from radiation to the lungs. The researchers hope that this study will help them in the future to design radiation treatment plans that provide the best treatment for each individual patient.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths in the United States, of which 80% are lung cancer (NSCLC, including squamous cell lung cancer, and small cell lung cancer). Although surgery provides the best chance of cure, the majority of lung cancer require radiation for treatment. The current radiation recommendation, using modern techniques and a uniform radiation dose, generates an overall cure rate of less than 10-15%, and moderate toxicity in 10-30% of treated patients. Who can be cured and who will develop side effects? Computed tomography (CT) provides a useful tool to monitor, but a limited power to predict both tumor control and lung toxicity. Using [18F] fluorodeoxyglucose positron emission tomography (FDG-PET) and ventilation/perfusion single photon emission computed tomography (V/Q SPECT), we have recently shown changes in tumor activity and regional lung function during the course of radiation, which may be associated with long-term outcome. The general strategy of this project is to perform functional image and blood test during the course of radiation and correlate them with long-term outcomes. By completing this study, we expect to generate predictive models better than CT-based ones for both tumor control and lung toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Non Small Cell Lung Cancer (NSCLC) or Small Cell Lung Cancer (SCLC) clinically diagnosed providing that FDG-PET is positive.
* Stage I to III lung cancer requiring definitive irradiation with or without chemotherapy.
* Patients with a locoregional tumor recurrence following surgery will be eligible provided they meet other eligibility criteria.
* Patients must be 18 years of age or older.
* Female patients with reproductive capability must be willing to use effective contraception
* Patients must sign an informed consent form for study.

Exclusion Criteria:

* Malignant pleural or pericardial effusion.
* Pregnancy
* Lactation
* Patients with diabetes mellitus, with uncontrolled fasting blood glucose level (above 200 mg/dl)
* Inability to lie flat for the duration of PET/CT and V/Q SPECT (approximately 45 minutes for each study)
* Prisoners are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2007-05; Primary Completion 2013-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study is to investigate predictive models for long-term tumor control and late treatment lung toxicity by using FDG-PET-CT, V/Q SPECT-CT and blood tests during the course of radiation therapy. | During treatment with radiation at 40-50 Gy and up to 5 yrs after radiation completed

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States